CLINICAL TRIAL: NCT04057261
Title: Effect of Liraglutide on the Metabolic Profile in Patients With Type 2 Diabetes and Cardiovascular Disease
Acronym: Lirabolic
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: A study start is currently not foreseeable for organizational reasons. Due to the delays, research has also been focused on new compounds, which has reduced the interest in the potential results of the above-mentioned clinical trial.
Sponsor: RWTH Aachen University (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 17-162
Record Dates: First submitted 2019-07-18; First posted 2019-08-15 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Type 2 Diabetes; Cardiovascular Diseases
Keywords: Liraglutide; Type 2 Diabetes; High Cardiovascular Risk; Myocardial Infarction; Metabolic Profile
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases; Myocardial Infarction | interventions — Liraglutide

STUDY DESIGN:
Intervention Model Description: Single center, prospective, placebo-controlled, double-blind, randomized, 2 arm parallel, interventional, exploratory pilot study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liraglutide (Active Comparator): Increasing dose of Liraglutide: 0.6 mg/d for the first week, 1.2 mg/d for the second week aiming for a maximum of 1.8 mg/d beginning with the third week (or highest tolerated dose).Subcutaneous injection once daily via pre-filled pen.
  Interventions: Drug: Liraglutide Pen Injector [Victoza]
- Placebo (Placebo Comparator): Matching Placebo once daily, subcutaneous injection via pre-filled pen.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Liraglutide Pen Injector [Victoza] — Increasing dose of Liraglutide: 0.6 mg/d for the first week, 1.2 mg/d for the second week aiming for a maximum of 1.8 mg/d beginning with the third week (or highest tolerated dose).Subcutaneous injection once daily via pre-filled pen
  Arms: Liraglutide
Drug: Placebo — Matching Placebo once daily, subcutaneous injection via pre-filled pen.
  Arms: Placebo

SUMMARY:
In an unbiased metabolomics approach with subsequent pathway analyses, the current study seeks to examine the effect of Liraglutide treatment on the metabolic signature in treated patients as well as the effect of Liraglutide on various echocardiographic parameters of cardiac function and rhythm profile, thus paving the way for future research to explain the effects of Liraglutide on cardiovascular mortality and overall mortality in treated patients.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes
2. Serum levels of HbA1c ≥ 7,0%
3. Age ≥ 18 years
4. Patients with existing cardiovascular disease: coronary heart disease, cerebrovascular disease, peripheral vascular disease, chronic kidney disease of stage III or chronic heart failure of NYHA II or III)
5. Written informed consent prior to study participation

Exclusion Criteria:

1. Type 1 diabetes
2. Treatment with GLP-1 receptor agonists or DPP-4 inhibitors within the last 4 weeks
3. Patients with familiar or personal history of multiple endocrine neoplasia-type 2 or medullary C-cell cancer
4. Renal impairment (eGFR < 30 mL/min)
5. Occurrence of acute vascular events within 6 weeks before screening and randomization
6. Known or suspected hypersensitivity to Liraglutide
7. Pregnant females as determined by positive (serum or urine) hCG test at Screening or prior to dosing. Participants of child-bearing age should use adequate contraception as defined in the study protocol.
8. Lactating females
9. The subject has a history of any other illness, which, in the opinion of the Investigator, might pose an unacceptable risk by administering study medication.
10. The subject received an investigational drug within 30 days prior to inclusion into this study.
11. The subject has any current or past medical condition and/or required medication to treat a condition that could affect the evaluation of the study.
12. The subject is unwilling or unable to follow the procedures outlined in the protocol.
13. The subject is mentally or legally incapacitated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-11 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Changes in the metabolomics profile (fold changes) between Liraglutide treatment group and placebo group after 1 and 3 months | 3 month
  Changes in the metabolomics profile (fold changes) between Liraglutide treatment group and placebo group after 1 and 3 months measured by a platform including 2 separate reverse phase (RP)/UPLC-MS/MS with positive ion mode electrospray ionization (ESI), (RP)/UPLC-MS/MS with negative ESI, and (HILIC)/UPLC-MS/MS with negative ESI.

SECONDARY OUTCOMES:
change in left ventricular diastolic function | 3 month
  change in left ventricular diastolic function between baseline and after 12 weeks as determined by 2D and 3D parameter global Strain Rate E by echocardiography
change in left ventricular diastolic function | 3 month
  change in left ventricular diastolic function between baseline and after 12 weeks as determined by standardized parameter E/é and left atrial (LA) volume by echocardiography
change in left ventricular systolic function | 3 month
  change in left ventricular systolic function by ejection fraction (EF) by echocardiography
Changes in systolic and diastolic blood pressure (mmHg) | 3 month
  Changes in systolic and diastolic blood pressure (mmHg) between Liraglutide treatment group and placebo group after 1 and 3 months.
body weight | 3 month
Changes in NT-proBNP serum levels (pg/ml) | 3 month
  Changes in NT-proBNP serum levels (pg/ml) between Liraglutide treatment group versus placebo group after 1 and 3 months.
Differences of the serum lipid profile between Liraglutide treatment group and placebo group | 3 month
  Differences of the serum lipid profile including serum levels of triglycerides (mg/dl), total cholesterol (mg/dl), low-density lipoprotein cholesterol (mg/dl) and high-density lipoprotein cholesterol (mg/dl)between Liraglutide treatment group and placebo group after 1 and 3 months
changes of serum levels of glucose, HbA1c, glucagon, insulin, C-Peptide, β-Hydroxybutyrate between Liraglutide treatment group and placebo group | 3 month
  Changes in serum levels of glucose (mg/dl), HbA1c (%), glucagon (pg/ml), insulin (ng/ml), C-Peptide (ng/ml), β-Hydroxybutyrate (mmol/l) between Liraglutide treatment group and placebo group after 1 and 3 months
Heart rate variability | 3 month
  Differences in heart rate variability measured by 24 hour ECG between Liraglutide treatment group and placebo group after 3 month including the following parameters: mean heart rate (bpm), maximum/minimum heart rate (bpm) and long-term variation of RR intervals (defined as standard deviation over 24 hours of per-minute means of RR intervals).
Resting energy expenditure | 3 month
  Resting energy expenditure measured by indirect calorimetry [CardioCoach CO2]
Respiratory Exchange Ratio | 3 month
  Respiratory Exchange Ratio measured by indirect calorimetry [CardioCoach CO2]
Differences in gut microbiome composition measured by 16S rRNA targeted gene sequencing of feces between Liraglutide treatment group and placebo group | 3 month
  Differences in gut microbiome composition measured by 16S rRNA targeted gene sequencing of feces between Liraglutide treatment group and placebo group after 1 and 3 month including the following parameters: alpha diversity (reported as Shannon diversity index) and differences in bacterial composition at different taxonomic levels including genus, family and class of bacteria (reported as relative abundance).
Albumin excretion | 3 month
  Albumin excretion by 24 h urine collection
changes in inflammasome analyses | 3 month
  Differences in serum levels of inflammatory cytokines including C-reactive protein (mg/ml), Interleukin 6 (pg/ml), Interleukin 1 beta (pg/ml) and tumor necrosis factor alpha (pg/ml) between Liraglutide treatment group and placebo group after 1 and 3 month
Differences in circulation inflammatory cell composition by flow cytometry analyses (FACS) between Liraglutide treatment group and placebo group | 3 month
  Differences in circulation inflammatory cell composition by flow cytometry analyses (FACS) between Liraglutide treatment group and placebo group after 1 and 3 month including the following parameters: Numbers of T-cells including T-cell subsets and monocytes including monocyte subsets. Numbers will be reported as percentage of parent, i.e. total pool of CD45+ immune cells).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine I, University Hospital, Aachen, Germany